CLINICAL TRIAL: NCT01682954
Title: Evaluation of a Lifestyle Intervention for Employees With Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Carla Miller, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012H0149; 1R34DK093907 (NIH)
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Prediabetes; Overweight; Obese
Keywords: lifestyle risk reduction
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): Diabetes Prevention Program lifestyle intervention
  Interventions: Behavioral: Lifestyle counseling
- Usual Care (No Intervention): Usual care from primary care physician

INTERVENTIONS:
Behavioral: Lifestyle counseling — 16-week nutrition, physical activity and behavioral intervention
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study is to evaluate the impact of a worksite lifestyle intervention for diabetes prevention among employees with prediabetes.

DETAILED DESCRIPTION:
The lifestyle intervention includes a 16-week group-based program which targets weight reduction through the adoption of a lower fat diet and greater physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* overweight or obese
* prediabetes with elevated glucose value

Exclusion Criteria:

* recent cardiovascular event
* use of corticosteroids
* concurrent participation in a structured weight loss program
* pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Miller, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Weinhold KR, Miller CK, Marrero DG, Nagaraja HN, Focht BC, Gascon GM. A Randomized Controlled Trial Translating the Diabetes Prevention Program to a University Worksite, Ohio, 2012-2014. Prev Chronic Dis. 2015 Nov 25;12:E210. doi: 10.5888/pcd12.150301. PMID 26605710
- [Derived] Miller CK, Nagaraja HN, Weinhold KR. Early weight-loss success identifies nonresponders after a lifestyle intervention in a worksite diabetes prevention trial. J Acad Nutr Diet. 2015 Sep;115(9):1464-71. doi: 10.1016/j.jand.2015.04.022. Epub 2015 Jun 19. PMID 26095435
- [Derived] Miller CK, Weinhold K, Marrero DG, Nagaraja HN, Focht BC. A Translational Worksite Diabetes Prevention Trial Improves Psychosocial Status, Dietary Intake, and Step Counts among Employees with Prediabetes: A Randomized Controlled Trial. Prev Med Rep. 2015;2:118-126. doi: 10.1016/j.pmedr.2015.02.003. PMID 25798374

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle Counseling | Usual Care
Started | 40 | 38
Completed | 35 | 33
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Counseling | Usual Care | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.75 (9.49) | 50.55 (7.99) | 50.65 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 40 | 38 | 78

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Change in body weight
Time Frame: 4 months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 35 | 34
kg | -5.12 (0.63) | -0.37 (0.64)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs Usual Care; Test type: Superiority or Other; p < 0.0001, ANOVA

2. Primary Outcome: Body Weight
Description: Change in body weight
Time Frame: 7 Months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Lifestyle Counseling | Usual Care
Number analyzed (Participants) | 35 | 33
kg | -4.86 (0.62) | -0.35 (0.64)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs Usual Care; Test type: Superiority or Other; p < 0.0001, ANOVA

ADVERSE EVENTS:
Arm/Group | Lifestyle Counseling | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 0/40 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No